CLINICAL TRIAL: NCT00990847
Title: The Efficacy of Nebulized Procaterol Versus Nebulized Salbutamol for the Treatment of Moderate Acute Asthma: a Randomized, Double-blind, Parallel Group Study
Brief Title: Nebulized Procaterol Versus Nebule Salbutamol for the Treatment of Moderate Acute Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PT Otsuka Indonesia (Industry)
Responsible Party: Albertus Widjaja/Medical Director, PT Otsuka Indonesia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 002-IOA-0601
Record Dates: First submitted 2009-10-05; First posted 2009-10-07 (Estimated); Last update posted 2009-10-07 (Estimated); Status verified 2009-10

CONDITIONS: Moderate Acute Asthma
MeSH Terms: interventions — Procaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Procaterol (Experimental): Procaterol inhalation solution 50 micro g per 0.5 mL diluted in 2mL of NaCl 0.9%, so that the volume of the inhalation solution will be similar to that of the comparator drug. The nebule solution will be administered 3 times, i.e. at times 0, 20 and 40 minutes.
  Interventions: Drug: Procaterol, Salbultamol
- Salbultamol (Active Comparator): Salbultamol inhalation solution for nebulization containing 2.5 mg in 2.5 mL aqueous solution. The nebule solution will be administered 3 times, i.e. at times 0, 20 and 40 minutes.
  Interventions: Drug: Procaterol, Salbultamol

INTERVENTIONS:
Drug: Procaterol, Salbultamol

SUMMARY:
The purpose of this study is to compare the efficacy and safety of nebule procaterol with nebule salbutamol in the treatment of moderate acute asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with moderate acute asthma according to Global Initiative for Asthma (GINA) 1998 (Appendix 1). Patients with moderate acute asthma according to Modified Global Initiative for Asthma (GINA) 1998 (Patients with asthma score 5 - 11; PEFR ≤ 80% predicted)
2. Patients of both gender aged 15 to 60 years
3. Patients still have the ability to undergo examinations and give written informed consent

Exclusion Criteria:

1. Pregnant and lactating women
2. Smokers
3. Patients with heart disease, hyperthyroidism, diabetes mellitus, COPD or other chronic diseases
4. Patients with signs of severe infections

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Difference 5% from baseline in peak expiratory flow rate (PEFR) | 3 times every 20 minutes (at 0, 20 and 40 minutes)

SECONDARY OUTCOMES:
Difference 5% from baseline in asthma score | 3 times every 20 minutes (at 0, 20 and 40 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Hadiarto Mangunnegoro, MD, Principal Investigator — Department of Pulmonology and Respiratory Medicine, Faculty of Medicine University of Indonesia/ Persahabatan Hospital
Locations (1):
- University of Indonesia/ Persahabatan Hospital, Jakarta, Indonesia